CLINICAL TRIAL: NCT00529906
Title: Endophenotype, Molecular Genetic Study on Attention-deficit/ Hyperactivity Disorder
Brief Title: Endophenotype, Molecular Genetic Study on Attention-Deficit/Hyperactivity Disorder
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Science and Technology Council, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 200612114R
Record Dates: First submitted 2007-09-13; First posted 2007-09-14 (Estimated); Last update posted 2021-05-07 (Actual); Status verified 2009-12

CONDITIONS: Attention Deficit Hyperactivity Disorder
Keywords: attention deficit hyperactivity disorder; neuropsychological deficits; endophenotype; molecular genetics; candidate gene; family-based association study
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Other
Biospecimen Retention: Samples With DNA — The subjects will receive blood withdrawal. The blood sample will be used for establishing lymphoblastoid cell lines, which will be used for molecular genetic experiments
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The ultimate goals of this study are to identify patterns of familial aggregation with regards to categorical and dimensional approaches of ADHD and neuropsychological measures, to validate the phenotypes and endophenotypes that are close to biological expression of genders underlying ADHD, and to identify the genetic variants close to the etiological genes of ADHD in Taiwanese sample. We propose to replicate the analysis of the candidate genes identified by previous genetic studies on ADHD using the candidate gene association study design (family-based case control study using parental controls) to validate the findings from other research groups. With the accomplishment of these goals, this study will resolve controversies over inconsistent findings in previous genetic studies and contribute to the literature on the validity of ASD using clinical and genetic data.

DETAILED DESCRIPTION:
Attention deficit hyperactivity disorder (ADHD), characterized by inattention, hyperactivity and impulsivity, is an early onset, highly heritable, clinically heterogeneous, long-term impairing disorder with tremendous impact on individuals, families, and societies. It affects 5-10% of school-aged children worldwide (7.5% in Taiwan) and 2-4% of adults. Neuropsychological deficits related to executive functions, state regulation, and delay aversion show heritability, replicated association with ADHD, and familial-genetic overlap with ADHD, are suitable for biomarkers for ADHD. Despite the abundance of molecular genetic studies on ADHD, the genetic etiologies of ADHD have been non-conclusive, and there is limited information about the expressions, endophenotypes, and genetic variants for ADHD in Chinese population. This polite study, a family-based parental control association study, aims to identify the genetic markers for ADHD using the dichotomous categorization of affected and non-affected, quantitative phenotypes (symptoms dimension and severity of ADHD) and endophenotype (neuropsychological measures) as well.

Specific Aims:

1. to determine the components of ADHD and neuropsychological deficit with the greatest familial recurrence risks;
2. to replicate studies with positive genetic findings from literature by performing candidate gene analysis such as DRD4, DAT1, DRD5, HTR1B, SNPA-25, 5-HTT, DBH, CHRNA4, CHRNA7 etc;
3. to identify the potential genetic variants using haplotype tag SNPs for the following candidate genes, CHRNA4 and CHRNA7 and any updated genetic findings.

We will recruit 200 probands with ADHD, aged 7-18, and their parents (n = 400) and siblings (n= 150) in three years (50, 100, and 50 families with ADHD in the 1st, 2nd, and 3rd year, respectively). The measures include (1) interviews for psychopathology (K-SADS-E) and social functioning (SAICA), (2) self-administered questionnaires to measures ADHD symptoms (CPRS-R:S, CTRS-R:S, SNAP-IV and Adult ADHD rating scale) and comorbid conditions (ASRI and CBCL), and (3) Neuropsychological tests: WISC-III, CPT, CANTAB, and Time Perception Tasks. The DNA will be collected and analyzed. The transmission/disequilibrium test (TDT) and quantitative TDT will be used in data analysis.

We anticipate the establishment of clinical, neuropsychological, and genetic database of 200 ADHD families, completion of the screening of several candidate genes, and identification of potential genetic variants for ADHD, and determination of their association with ADHD diagnosis and symptoms and its endophenotype in a Taiwanese sample. The long-term objectives are to identify the behavioral phenotypes and endophenotypes that are close to the biological expression of genes underlying ADHD. The findings of different approaches to identify the genetic etiologies for ADHD in this pilot study should help us to determine the most promising approach for future molecular genetic study on ADHD.

ELIGIBILITY:
Inclusion Criteria:

The inclusion criteria for the proband subjects are

* (1) that subjects have a clinical diagnosis of ADHD, or Hyperkinetic Disorder (HD) defined by the DSM-IV and ICD-10, respectively, which was made by a full-time board-certificated child psychiatrist at the first visit and following visits;
* (2) their ages range from 7 to 18 when we conduct the study;
* (3) subjects have at least one biological parent;
* (4) both parents are Han Chinese; and
* (5) subjects and their biological parents (and siblings if any) consent to participate in this study for complete phenotype assessments and blood withdraw or saliva collection for genetic study

Exclusion Criteria:

* The proband subjects will be excluded from the study if they currently meet criteria or have a history of the following condition as defined by DSM-IV:
* Shizophrenia,
* Schizoaffective Disorder,
* Organic Psychosis, or Pervasive Developmental Disorder.
* Moreover, the subjects will also be excluded from the study if they completely cannot cooperate with blood withdrawal, collection of saliva, or buccal swabs.

Ages: 7 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The sample will consist of 200 children and adolescents with ADHD, aged 7-18.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2007-08; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Shur-Fen Gau, MD, PhD, Principal Investigator — Dept of Psychiatry, National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Chiang HL, Gau SS. Impact of executive functions on school and peer functions in youths with ADHD. Res Dev Disabil. 2014 May;35(5):963-72. doi: 10.1016/j.ridd.2014.02.010. Epub 2014 Mar 11. PMID 24636025
- [Derived] Gau SS, Chiang HL. Association between early attention-deficit/hyperactivity symptoms and current verbal and visuo-spatial short-term memory. Res Dev Disabil. 2013 Jan;34(1):710-20. doi: 10.1016/j.ridd.2012.10.005. Epub 2012 Nov 5. PMID 23137723